CLINICAL TRIAL: NCT01582191
Title: A Phase 1 Trial of Vandetanib (a Multi-Kinase Inhibitor of EGFR, VEGFR, and RET Inhibitor) in Combination With Everolimus (an mTOR Inhibitor) in Advanced Cancer
Brief Title: Vandetanib and Everolimus in Treating Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0953; NCI-2012-00782 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0953; 2011-0953 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Neoplasm; Metastatic Malignant Neoplasm; Recurrent Malignant Neoplasm; Refractory Malignant Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Recurrence; Neoplasms | interventions — Everolimus; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (vandetanib, everolimus) (Experimental): Patients receive vandetanib PO QD and everolimus PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Everolimus; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Vandetanib

INTERVENTIONS:
Drug: Everolimus — Given PO
  Other Names: 42-O-(2-Hydroxy)ethyl Rapamycin; Afinitor; Certican; RAD 001; RAD001; Votubia; Zortress
Other: Laboratory Biomarker Analysis — Optional correlative studies
Other: Pharmacological Study — Optional correlative studies
Drug: Vandetanib — Given PO
  Other Names: AZD6474; Caprelsa; Zactima; ZD-6474; ZD6474

SUMMARY:
This phase I trial studies the side effects and best dose of vandetanib and everolimus when given together in treating patients with cancer that has spread to other places in the body. Vandetanib and everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) or highest dose level, and the dose-limiting toxicity (DLT) of vandetanib (a multi-kinase inhibitor of epidermal growth factor receptor [EGFR], vascular endothelial growth factor receptor [VEGFR] and ret proto-oncogene [RET] inhibitor) when used in combination with everolimus (a mammalian target of rapamycin [mTOR] inhibitor) in advanced cancer.

II. Preliminary descriptive assessment of the anti-tumor efficacy of the combination.

III. Preliminary optional assessment of the pharmacokinetic, pharmacodynamic markers of target inhibition and correlates of response.

OUTLINE: This is a dose-escalation study.

Patients receive vandetanib orally (PO) once daily (QD) and everolimus PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment patients are followed up between 14-28 days at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic cancer that is refractory to standard therapy, relapsed after standard therapy, or who have no standard therapy available that improves survival by at least three months.
* Patients must be at least 3 weeks beyond their previous cytotoxic chemotherapy.
* Patient must be at least 5 half-lives or 3 weeks, whichever is shorter, from their previous targeted or biologic therapy; In addition, patients must be at least 3 weeks beyond the last session of radiation therapy. Local palliative radiation therapy that is not delivered to all target lesions is allowed immediately before or during treatment.
* ECOG performance status should be less or equal to 3
* Patients must have organ and marrow function defined as: Absolute neutrophil count more or equal to 750/mL; platelets more or equal to 50,000/mL; creatinine less or equal to 3x ULN; total bilirubin less than or equal to 3.0.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence).

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, uncontrolled asthma, need for hemodialysis, need for ventilatory support.
* Pregnant or lactating women.
* History of hypersensitivity to vandetanib, lactose, murine products, or any component of the formulation.
* History of hypersensitivity to sirolimus, temsirolimus, everolimus.
* History of hypersensitivity to any component of the formulation.
* Patients unwilling or unable to sign informed consent document.
* Presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* History (within the last 3 months) or presence of stroke/cerebrovascular accident.
* Congenital long QT syndrome.
* QTcF interval greater than 500 ms that is not correctable to less than 500ms such as with cessation of a causative medication, etc.
* History of myocardial infarction within 6 months with a residual arrhythmia that in the opinion of the Investigator, increases the risk of ventricular arrhythmia.
* Presence of a symptomatic bradyarrhthmia or uncompensated heart failure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2012-05-14 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 28 days
  Will be defined as the highest dose studied in which the incidence of dose limiting toxicity was less than 33%. Toxicity will be reported by type, frequency, and severity. Worst toxicity grades per patient will be tabulated for selected adverse events and laboratory measurements.
Anti-tumor efficacy of the combination in terms of response rate | Up to 14 years
  The response rate will be estimated by dose level and tumor type, along with the exact 95% confidence interval. Efficacy will be evaluated by using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria described in the supplement for response. Patients with lymphoma will be measured per the World Health Organization (WHO) criteria.
Maximum observed serum concentration (Cmax) | Days 1 and 21 of course 1 and day 1 of course 3
  Will be estimated using standard non-compartmental methods
Pharmacodynamic (PD) parameters | Up to 14 years
  PD biomarker concentration will be summarized by time points. The relationship between drug concentrations and PD effects will be explored graphically. Based on review of these graphs, analyses to describe the relationship may also be performed.
Observed trough serum concentration (Cmin) | Days 1 and 21 of course 1 and day 1 of course 3
  Will be estimated using standard non-compartmental methods
Area under the serum concentration-time curve (AUC) | Days 1 and 21 of course 1 and day 1 of course 3
  Will be estimated using standard non-compartmental methods

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Piha-Paul, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Subbiah V, Berry J, Roxas M, Guha-Thakurta N, Subbiah IM, Ali SM, McMahon C, Miller V, Cascone T, Pai S, Tang Z, Heymach JV. Systemic and CNS activity of the RET inhibitor vandetanib combined with the mTOR inhibitor everolimus in KIF5B-RET re-arranged non-small cell lung cancer with brain metastases. Lung Cancer. 2015 Jul;89(1):76-9. doi: 10.1016/j.lungcan.2015.04.004. Epub 2015 Apr 22. PMID 25982012
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT01582191/ICF_000.pdf